CLINICAL TRIAL: NCT06630156
Title: Clinical and Radiographic Evaluation of Bioceramic Root Repair Versus Bio MTA in Revascularization of Immature Young Permenant Teeth.
Brief Title: The Present Study Was Conducted to Evaluate Bioceramic Root Repair Material Versus Bio MTA in Revascularization of Immature Young Permenant Teeth.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Reda Mohammed Mohammed Elsayed, assistant lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Treatment of immature teeth
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Revascularization of Immature Young Permenant Teeth
Keywords: Revascularization; Bio MTA; Total Fill biocearmic root repair material

STUDY DESIGN:
Intervention Model Description: The patients selected in this study were randomly divided into 2 groups:
  1. Group A: 14 teeth were disinfected by triple paste and treated by Bio-MTA.
  2. Group A: 14 teeth were disinfected by triple paste and treated by a Total Fill biocearmic root repair.
Who Masked: Participant, Outcomes Assessor
Masking Description: The statistician and the assessor were blinded, but the operator was not because of the nature of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bio-MTA revascularization (Active Comparator)
  Interventions: Biological: Revascularization of Immature Young Permenant Teeth
- Total Fill biocearmic root repair material revascularization (Active Comparator)
  Interventions: Biological: Revascularization of Immature Young Permenant Teeth

INTERVENTIONS:
Biological: Revascularization of Immature Young Permenant Teeth — An access cavity was prepared under rubber dam, isolation, root canal system disinfection was done without mechanical instrumentation. Subsequently, triple antibiotic paste was placed into the apical portion of the canal and filled to just below the CEJ. The access cavity was temporarily restored with glass ionomer.
  4 weeks later, after reopening of the access, the antibiotic paste was gently flushed out of the canal with sterile normal saline. The root canal system was irrigated. A sterile #35 K-file will be introduced into the canal beyond the apical foramen using a push and pull motion to provoke bleeding from the periapical tissue. After bleeding control and formation of fresh blood clot, 3 mm of Bio (MTA) will be placed in Group A, 3 mm of Total Fill biocearmic root repair material will be placed in Group B after a moist cotton pellet was placed over the capping material and the access cavity will be sealed with G C

SUMMARY:
The present clinical study wasdirected to evaluate bioceramic root repair material versus Bio MTA in Revascularization of Immature Young Permenant Teeth through:

1. Clinical evaluation including: Pain, swelling, sinus or fistula, mobility and crown discoloration.
2. Radiographic evaluation including: Root lengthening, continued thickening of the dentinal walls, apical closure and regression of the peri-apical lesion.

DETAILED DESCRIPTION:
In a young permanent tooth with pulp necrosis and apical pathosis, routine endodontic treatment may not be possible due to the immature apex it possesses. Newer methods based on the principles of revascularization and regeneration have been tried and found to be much better than the traditional methods of apexification since it helps in physiological root maturation, unlike traditional methods which result in only artificial barrier formation without root lengthening.

Revascularization is a new treatment method for immature necrotic permanent teeth. Indeed, it would provide, after treatment, a vital tooth that would be able to complete its root maturation. Three key requirements for a successful revascularization are: (a) Root canal disinfection; (b) matrix inside the canal for growth of tissue (scaffold); and (c) a tight seal access filling.

Bio MTA was introduced to overcome some of the drawbacks of MTA such as handling properties and long setting time. Bio MTA has a faster setting time with good handling characteristics and biological properties. Calcium silicate based restorative cements were formulated using different calcium compounds such as calcium hydroxide, calcium oxide, calcium phosphate, calcium sulfate, calcium silicate, and calcium carbonate in combination with zirconium. The mixed cement comprises water-soluble calcium and phosphate and immediately forms hydroxyapatite during and after setting.

A Total Fill biocearmic root repair material which is calcium silicate-based cement was developed with excellent handling properties as it is supplied in premixed packages (putty) that do not require preparation before use. It is mainly composed of calcium silicate, monobasic calcium phosphate, calcium hydroxide, and zirconium oxide. It has antibacterial and antifungal activities. It is claimed that the material is biocompatible with human periodontal tissues.

ELIGIBILITY:
Inclusion Criteria:

1. Child with an age ranged from (7-12) year from both sexes.
2. Patient and parent cooperation.
3. Non vital immature permanent teeth indicated for endodontic treatment as a result of pulp necrosis.
4. Patient is not taking antibiotic and has not taken for the past 2 weeks.
5. Restorable teeth.
6. The root to crown ratio should be at least 1:1.

Exclusion Criteria:

1. Patients allergic to any drug used in this RCT.
2. Patients with any systemic disease that would contraindicate pulp therapy (rheumatic fever, infective endocarditis, leukemia, corticosteroid therapy and immune suppressed children).
3. Tooth with vital pulp or complete root formation.
4. Teeth with draining sinus or periodontal weak mobile teeth.
5. Teeth with internal or external root resorption.
6. Tooth with root fracture.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2022-08-21 (Actual); Primary Completion 2024-11-21 (Estimated); Study Completion 2024-12-21 (Estimated)

PRIMARY OUTCOMES:
radiographic parameters | baseline, 3, 6, and 12 months after treatment
  continued root lengthening and thickening of the dentinal walls in mm

CONTACTS AND LOCATIONS:
Overall Officials: Reda Mohammed Elsayed, assistant lecturer, Principal Investigator — Faculty of Dental Medicine, Al- Azhar University, Assuit, Egypt
Locations (1):
- faculty of dental medicine, Al-Azhar university, Asyut, Egypt

REFERENCES:
- [Background] Murray PE, Garcia-Godoy F, Hargreaves KM. Regenerative endodontics: a review of current status and a call for action. J Endod. 2007 Apr;33(4):377-90. doi: 10.1016/j.joen.2006.09.013. Epub 2007 Feb 20. PMID 17368324
- [Background] Kim DS, Park HJ, Yeom JH, Seo JS, Ryu GJ, Park KH, Shin SI, Kim SY. Long-term follow-ups of revascularized immature necrotic teeth: three case reports. Int J Oral Sci. 2012 Jun;4(2):109-13. doi: 10.1038/ijos.2012.23. PMID 22627612
- [Background] Bose R, Nummikoski P, Hargreaves K. A retrospective evaluation of radiographic outcomes in immature teeth with necrotic root canal systems treated with regenerative endodontic procedures. J Endod. 2009 Oct;35(10):1343-9. doi: 10.1016/j.joen.2009.06.021. Epub 2009 Aug 15. PMID 19801227
- [Background] Shuping GB, Orstavik D, Sigurdsson A, Trope M. Reduction of intracanal bacteria using nickel-titanium rotary instrumentation and various medications. J Endod. 2000 Dec;26(12):751-5. doi: 10.1097/00004770-200012000-00022. PMID 11471648
- [Background] Chen MY, Chen KL, Chen CA, Tayebaty F, Rosenberg PA, Lin LM. Responses of immature permanent teeth with infected necrotic pulp tissue and apical periodontitis/abscess to revascularization procedures. Int Endod J. 2012 Mar;45(3):294-305. doi: 10.1111/j.1365-2591.2011.01978.x. Epub 2011 Nov 14. PMID 22077958
- [Background] Asgary S, Fazlyab M, Nosrat A. Regenerative Endodontic Treatment versus Apical Plug in Immature Teeth: Three-Year Follow-Up. J Clin Pediatr Dent. 2016;40(5):356-60. doi: 10.17796/1053-4628-40.5.356. PMID 27617375
- [Background] Chuensombat S, Khemaleelakul S, Chattipakorn S, Srisuwan T. Cytotoxic effects and antibacterial efficacy of a 3-antibiotic combination: an in vitro study. J Endod. 2013 Jun;39(6):813-9. doi: 10.1016/j.joen.2012.11.041. Epub 2013 Jan 27. PMID 23683284
- [Background] Banchs F, Trope M. Revascularization of immature permanent teeth with apical periodontitis: new treatment protocol? J Endod. 2004 Apr;30(4):196-200. doi: 10.1097/00004770-200404000-00003. PMID 15085044
- [Background] Jitaru S, Hodisan I, Timis L, Lucian A, Bud M. The use of bioceramics in endodontics - literature review. Clujul Med. 2016;89(4):470-473. doi: 10.15386/cjmed-612. Epub 2016 Oct 20. PMID 27857514
- [Background] Alobaid AS, Cortes LM, Lo J, Nguyen TT, Albert J, Abu-Melha AS, Lin LM, Gibbs JL. Radiographic and clinical outcomes of the treatment of immature permanent teeth by revascularization or apexification: a pilot retrospective cohort study. J Endod. 2014 Aug;40(8):1063-70. doi: 10.1016/j.joen.2014.02.016. Epub 2014 Jun 13. PMID 25069909
- [Background] Torabinejad M, Pitt Ford TR. Root end filling materials: a review. Endod Dent Traumatol. 1996 Aug;12(4):161-78. doi: 10.1111/j.1600-9657.1996.tb00510.x. PMID 9028180